CLINICAL TRIAL: NCT02556996
Title: Efficacy of an Oral, Killed Enterotoxigenic Escherichia Coli Vaccine in Prevention of Diarrhea in Egyptian Infants and Young Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: U.S. Naval Medical Research Unit No. 3 (Unknown); Ministry of Health and Population, Egypt (Other Government); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); International Vaccine Institute (Other); Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HSRRB A-7965
Record Dates: First submitted 2015-09-21; First posted 2015-09-22 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Diarrhea
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Killed ETEC/rCTB vaccine (Experimental): Three doses administered orally at 2-week intervals
  Interventions: Biological: ETEC/rCTB vaccine
- Placebo (Placebo Comparator): Three doses administered orally at 2-week intervals
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: ETEC/rCTB vaccine — Cocktail of five whole-cell, formalin-inactivated ETEC strains (total of 10^11 formalin-killed bacteria per dose) plus recombinant cholera toxin B-subunit (rCTB) (1 mg)
  Arms: Killed ETEC/rCTB vaccine
Other: Placebo — Heat-killed, nonpathogenic E. coli K-12 bacteria (total of 10^11 heat-killed bacteria per dose)
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled clinical trial performed in Egyptian children 6-18 months of age. The primary aim of the study is to determine the protective efficacy of an oral, inactivated whole-cell enterotoxigenic Escherichia coli (ETEC) vaccine against diarrhea associated with excretion of ETEC that express a vaccine-shared antigen over a one year period of follow-up by active surveillance. The vaccine consists of a mixture of five formalin-killed ETEC bacteria expressing prevalent ETEC colonization factors and recombinant cholera toxin B-subunit (killed ETEC/rCTB vaccine). The placebo preparation is heat-killed Escherichia coli K-12 bacteria.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness of parent to have the child participate;
2. Plans to reside in catchment area continuously for at least one year

Exclusion Criteria:

1. Global developmental delay
2. Severe malnutrition
3. Chronic bedridden status
4. Serious chronic disorder requiring chronic medication

Ages: 6 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 356 (Actual)
Dates: Start 1998-10; Primary Completion 2001-03 (Actual); Study Completion 2002-04 (Actual)

PRIMARY OUTCOMES:
Time to first event of diarrhea due to vaccine-preventable ETEC (VP-ETEC) as defined below, and no other copathogen. | 365-day period starting 14 days after the third vaccination
  Time to first event of diarrhea associated with excretion of VP-ETEC (defined as ETEC expressing heat-labile [LT] and heat-stable enterotoxin [ST], or ST and a vaccine-shared colonization factor [i.e., CFA/I, CS1, CS2, CS3, CS4, and/or CS5]) and no other copathogen.

SECONDARY OUTCOMES:
Time to first event of diarrhea due to ST-only ETEC expressing a vaccine-shared CF (ST-VCF-ETEC) as defined below, and no other copathogen.. | 365-day period starting 14 days after the third vaccination
  Time to first event of diarrhea associated with excretion of ST-VCF-ETEC (defined as ETEC expressing ST-only plus any vaccine-shared colonization factor [i.e., CFA/I, CS1, CS2, CS3, CS4, and/or CS5]) and no other copathogen.
All events of diarrhea irrespective of etiology | 365-day period starting 14 days after the third vaccination
  All events (i.e., initial plus recurrent) of diarrhea associated with excretion of any ETEC, irrespective of phenotype, and no other copathogen.
IgG seroconversion | Baseline serum specimen is collected before first dose and post-vaccination specimen collected 14 days after third dose
  IgG seroconversion (≥ twofold increase in post-vaccination endpoint titer over baseline) against rCTB and vaccine-specific colonization factors CFA/I, CS2, CS4
IgA seroconversion | Baseline serum specimen is collected before first dose and post-vaccination specimen collected 14 days after third dose
  IgA seroconversion (≥ twofold increase in post-vaccination endpoint titer over baseline) against rCTB and selected vaccine-specific colonization factors CFA/I, CS2, CS4
Number of solicited adverse events | 3-day period after each dose
  (i.e., diarrhea, vomiting, fever by caregiver report, poor feeding, and irritability)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Savarino, MD, MPH, Principal Investigator — Naval Medical Research Center